CLINICAL TRIAL: NCT00148772
Title: Phase II Study of Erlotinib in Patients With Non-Metastatic Prostate Cancer With a Rising PSA on Hormone Therapy
Brief Title: Study of Erlotinib in Patients With Non-Metastatic Prostate Cancer With a Rising Prostate Specific Antigen (PSA) on Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Genentech, Inc. (Industry); Northwestern University (Other)
Responsible Party: Daniel Shevrin, MD, NorthShore University HealthSystem
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSI3316s
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2005-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Rising PSA; Erlotinib; Tarceva; Androgen Deprivation Therapy; Hormone Therapy; Rising Prostate Specific Antigen (PSA); Non-Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Erlotinib (Tarceva)

SUMMARY:
The primary objective of this study is to evaluate the effect of erlotinib on the PSA response rate in patients with non-metastatic prostate cancer and a rising PSA on androgen deprivation therapy.

The secondary objectives are to evaluate the effect of erlotinib on the duration of PSA response, to evaluate the effect on the time to PSA progression, to evaluate the toxicity of erlotinib in this patient population, and lastly, to correlate the effect of erlotinib with various epidermal growth factor receptor (EGFR)-related proteins using baseline immunohistochemical (IHC) studies on tissue blocks and peripheral blood mononuclear cells.

DETAILED DESCRIPTION:
Patients with prostate cancer who are treated with surgery or radiation often develop recurrence of their cancer which is manifest only by a rising PSA (Prostate Specific Antigen) level. Many of these patients are treated with hormone therapy. After a fall in the PSA, these patients eventually display evidence of tumor progression clearly demonstrated by another rise in PSA level while receiving hormone therapy. Evaluation for evidence of tumor spread is usually negative. There is currently no effective therapy approved for use in these patients.

The drug erlotinib works by blocking the activity of a protein called Epidermal Growth Factor Receptor (EGFR), which is located on the surface of many prostate cancer cells. Blockage of this protein has been shown to inhibit the growth of prostate tumor cells in a laboratory setting and in animal experiments. Erlotinib has been given to patients with other types of cancers. A recently completed study showed that erlotinib improved the survival of patients with advanced lung cancer who failed standard chemotherapy.

There is currently no effective therapy approved for use in patients with this condition. The purpose of this study is to evaluate the effectiveness and side effects of the drug erlotinib in patients with this condition. Erlotinib is an investigational drug that has not yet been approved by the Federal Drug Administration (FDA) for use in prostate cancer, but has been approved for use in lung cancer.

As previously stated: The primary objective of this study is to evaluate the effect of erlotinib on the PSA response rate in patients with non-metastatic prostate cancer and a rising PSA on androgen deprivation therapy.

Secondary objectives are to evaluate the effect of erlotinib on the duration of PSA response, to evaluate the effect on the time to PSA progression, to evaluate the toxicity of erlotinib in this patient population, and lastly, to correlate the effect of erlotinib with various EGFR-related proteins using baseline immunohistochemical (IHC) studies on tissue blocks and peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documented adenocarcinoma of the prostate, treated with androgen suppression, and now present with a rising PSA .
* Prior therapy with hydrocortisone is allowed (must have discontinued > 4 weeks prior to study treatment). Prior use of ketoconazole for prostate cancer treatment is allowed (must have discontinued > 4 weeks prior to study treatment).
* Prior therapy with chemotherapy is allowed if it was administered as neoadjuvant or adjuvant therapy related to primary treatment and was completed > 6 months prior to starting study treatment.
* Testosterone level < 50 ng/dl within 4 weeks prior to study treatment. Patients who have not undergone surgical castration must continue primary androgen suppression therapy (luteinizing hormone-releasing hormone [LHRH] agonist) while on protocol therapy.
* Patients may be receiving oral bisphosphonate therapy prior to study treatment and continue while receiving treatment, but must not begin treatment with bisphosphonate while receiving study treatment. Patients on oral bisphosphonates must have completed at least 4 weeks of bisphosphonate therapy prior to study treatment.
* Patients must have adequate major organ function. All values must be obtained within 4 weeks prior to study treatment.

  * Creatinine < 1.7 mg/dL or a creatinine clearance > 50 mL/min,
  * SGOT (AST), SGPT (ALT) < 2X the institution's upper limit of normal,
  * Bilirubin < 1.5 mg/dL,
  * ANC > 1500/mm3,
  * Platelet (PLT) > 100,000/mm3
* Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Patients must be > 18.
* Patients taking warfarin are eligible.
* Patients taking CYP3A4 inducers or inhibitors are eligible.
* Patients with a history of prior malignancy are eligible provided they were treated with curative intent and have been free of disease for the time period considered appropriate for the specific cancer.

Exclusion Criteria:

* No previous palliative radiation. Prior radiation to the primary site is allowed.
* HIV positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with erlotinib.
* Patients with gastrointestinal tract disease resulting in an inability to take oral medication are ineligible.
* Patients must not have ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia, or psychiatric illness that would limit compliance with study requirements.
* Patients must not have received prior targeted therapy, including no prior EGFR inhibitor.
* Patients must not have evidence of metastatic disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2005-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of erlotinib on the PSA response rate in patients with non-metastatic prostate cancer and a rising PSA on androgen deprivation therapy

SECONDARY OUTCOMES:
To evaluate the effect of erlotinib on the duration of PSA response
To evaluate the effect of erlotinib on the time to PSA progression
To evaluate the toxicity of erlotinib in this patient population
To correlate the effect of erlotinib with various EGFR downstream proteins and androgen receptor, using baseline IHC studies on tissue blocks and analysis of protein phosphorylation in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Shevrin, MD, Principal Investigator — Endeavor Health
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois